CLINICAL TRIAL: NCT05320952
Title: Effect of Upper Respiratory Muscle Strength Exercise on Sleep Apnea Using WellO2 Respiratory Exercise Device
Brief Title: Muscle Strength Exercise and Sleep Apnea
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: WellO2 Oy (Industry); University of Turku (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TO5/004/22
Record Dates: First submitted 2022-02-24; First posted 2022-04-11 (Actual); Last update posted 2025-05-31 (Actual); Status verified 2025-05

CONDITIONS: Sleep Apnea
Keywords: sleep apnea; muscle strength exercise; WellO2; apnea hypopnea
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Intervention Model Description: Open label single group study with three months active phase followed by three months washout.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- working sleep apnea patients (Experimental): 50 sleep apnea patients with mild to moderate sleep apnea using WellO2 device for three months
  Interventions: Device: WellO2

INTERVENTIONS:
Device: WellO2 — The WellO2 breathing training device performs back-pressure steam breathing training during the inhalation and exhalation phases.

SUMMARY:
Background:

Obstructive sleep apnea is one of our common diseases and up to 80% of patients are estimated to be undiagnosed. Its main risk factors are overweight, age, male gender, menopause, small jaw, sedative medications / drugs and alcohol. The most important treatment for sleep apnea is continuous positive airway pressure (CPAP). However, not all patients adapt or benefit from device therapy, and up to about 60% stop using the device. Underlying sleep apnea are mechanisms other than anatomical factors such as respiratory wake sensitivity, loop gain control function, and upper respiratory tract muscle activation response and efficiency. Depending on which of these mechanisms dominates as the cause of sleep apnea, the patient's phenotype may vary and CPAP device therapy may not be the correct form of treatment for all patients. Therefore, new targeted therapies should be developed.

The WellO2 breathing training device performs back-pressure steam breathing training during the inhalation and exhalation phases. WellO2 effectively exercises the power of the inspiratory muscles, increases the inspiratory muscles, reduces the feeling of dyspnea due to exertion, increases the economy of respiration and delays inhalation muscles. It is a drug-free treatment and easy to use. The use of the WellO2 ventilator has not been previously studied in sleep apnea patients.

DETAILED DESCRIPTION:
Research objectives:

1. Will AHI change after 3 months of use of WellO2 (PSG in the beginning and after 3 months)
2. Will the participants get help with fatigue symptoms or quality of life (questionnaires)
3. Is there a response to WellO2 treatment in AHI and symptoms of sleep apnea still after 3 months of WellO2 treatment washout (PSG 3 months after treatment discontinuation)
4. Are the participants able to use the device (questionnaires)

Research design:

A clinical follow-up study in lung clinic sleep apnea patients who are not receiving any other form of sleep apnea treatment. The estimate for the recruitment phase is 6-12 months. The duration of the study is 6 months, of which the active phase with the WellO2 breathing apparatus is 3 months and the washout phase is 3 months after the end of treatment.

Material:

The study enrolled working sleep apnea patients aged 18 to 60 years (n = 50; M: N = 1: 1) with mild to moderate obstructive sleep apnea (AHI 10-29 / h). Exclusion criteria: Previous surgical treatment for sleep apnea, current CPAP or mandibular device therapy, significant history of nasal, oral and pharyngeal disorders, BMI> 40 kg / m2, other severe pulmonary diseases (eg COPD, asthma, pulmonary fibrosis) severe heart failure (NYHA 3-4), previous brain event, neuromuscular disease or pregnancy, and disability to work.

Methods:

Participants enrolled in the study will be selected from referrals coming to Turku University Hospital for pulmonary department due to sleep apnea. Participants are interviewed in a structured way and demographic and anthropometric data (gender, age, BMI, neck and waist circumference, smoking), sleep apnea symptoms, possible previous treatment attempts, and other known diseases and medications are collected from the interview and from the hospital's patient paper archive. Sleep apnea is examined by sleep polypomyography (polysomnography, PSG) at the beginning of the study, 3 months after WellO2 treatment, and 3 months after the end of treatment. Participants complete the following questionnaires: Epworth Sleepiness Scale (ESS), 12-item General Health Questionnaire (GHQ-12), Depression Survey (DEPS), Insomnia Severity Index (ISI), Pittsburgh Sleep Quality Index (PSQI), Sleep Apnea Symptom Survey, Satisfaction Survey. Measurements of maximal inspiratory pressure (MIP) and maximal expirium pressure (MEP) are used to assess muscle strength, and FEV1, FVC, FEV1 / FVC, and PEF are measured with a miniature spirometer to see the size of the large bronchi and possible bronchial obstruction.

The participant is instructed in the use of the WellO2 orally and in writing. The WellO2 device is used twice a day for 15 minutes at a time at a power corresponding to 30% of the participant's MEP / MIP value. The WellO2 comes with an accessory that records the times and times you have done, as well as the power with the help of a pressure sensor and a mobile assistant. The WellO2 device will continue to be used for a total of 3 months, followed by a second three-month follow-up period without the WellO2 device.

The primary endpoint is resolution of sleep apnea symptoms and PSG findings after 3 months of treatment. The secondary endpoint is whether the effect after 3 months of treatment is maintained after the next 3-month's washout phase.

Significance of the research:

The physiological causes of sleep apnea have been clarified thanks to research in recent years. Hyperbaric ventilator therapy is not suitable for everyone and new therapies are needed for these patients. So far, there is no cure for sleep apnea. The WellO2 breathing training device would be affordable and easy to use for properly targeted sleep apnea patients of all ages.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-60 years
* Male:Famel 1:1
* AHI 10-29 / h
* working patients

Exclusion Criteria:

* Previous surgical treatment for sleep apnea, current CPAP or mandibular device therapy
* significant history of nasal, oral and pharyngeal disorders
* BMI> 40 kg / m2
* other severe pulmonary diseases (eg COPD, asthma, pulmonary fibrosis) severe heart failure (NYHA 3-4), previous brain insult, neuromuscular disease or pregnancy, and work disability.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-23 (Actual); Primary Completion 2024-08-31 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Apnea-hypopnea index, AHI | 3 months
  Change in AHI measured from polysomnogaphy in the beginning and after 3 month's of WellO2 treatment?

SECONDARY OUTCOMES:
Sleep apnea symptoms | 3 months
  Is there a change in the sleep apnea symptoms (ex. fatigue symptoms or quality of life) after the WellO2 treatment?
Longterm benefits in AHI and symptoms of sleep apnea | 6 months
  Is there a change in AHI or sleep apnea symptoms due to the WellO2 treatment after 3 months of treatment washout?
WellO2 device usability | 3 months
  Are the participants able to use the WellO2 device during the 3 month's intervention?

CONTACTS AND LOCATIONS:
Overall Officials: Ulla Anttalainen, MD, PhD, Principal Investigator — Turku University Hospital, Turku, Finland
Locations (1):
- Turku University Hospital, Division of Medicine, Dept of Pulmonary diseases and University of Turku, Sleep Research Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Peppard PE, Young T, Barnet JH, Palta M, Hagen EW, Hla KM. Increased prevalence of sleep-disordered breathing in adults. Am J Epidemiol. 2013 May 1;177(9):1006-14. doi: 10.1093/aje/kws342. Epub 2013 Apr 14. PMID 23589584
- [Background] Afsharpaiman S, Shahverdi E, Vahedi E, Aqaee H. Continuous Positive Airway Pressure Compliance in Patients with Obstructive Sleep Apnea. Tanaffos. 2016;15(1):25-30. PMID 27403175
- [Background] Dempsey JA, Xie A, Patz DS, Wang D. Physiology in medicine: obstructive sleep apnea pathogenesis and treatment--considerations beyond airway anatomy. J Appl Physiol (1985). 2014 Jan 1;116(1):3-12. doi: 10.1152/japplphysiol.01054.2013. Epub 2013 Nov 7. PMID 24201709
- [Background] Eckert DJ. Phenotypic approaches to obstructive sleep apnoea - New pathways for targeted therapy. Sleep Med Rev. 2018 Feb;37:45-59. doi: 10.1016/j.smrv.2016.12.003. Epub 2016 Dec 18. PMID 28110857
- [Background] Enright SJ, Unnithan VB, Heward C, Withnall L, Davies DH. Effect of high-intensity inspiratory muscle training on lung volumes, diaphragm thickness, and exercise capacity in subjects who are healthy. Phys Ther. 2006 Mar;86(3):345-54. PMID 16506871
- [Background] Karsten M, Ribeiro GS, Esquivel MS, Matte DL. The effects of inspiratory muscle training with linear workload devices on the sports performance and cardiopulmonary function of athletes: A systematic review and meta-analysis. Phys Ther Sport. 2018 Nov;34:92-104. doi: 10.1016/j.ptsp.2018.09.004. Epub 2018 Sep 15. PMID 30261349
- [Background] Romer LM, McConnell AK. Specificity and reversibility of inspiratory muscle training. Med Sci Sports Exerc. 2003 Feb;35(2):237-44. doi: 10.1249/01.MSS.0000048642.58419.1E. PMID 12569211
- [Background] Romer LM, McConnell AK, Jones DA. Effects of inspiratory muscle training on time-trial performance in trained cyclists. J Sports Sci. 2002 Jul;20(7):547-62. doi: 10.1080/026404102760000053. PMID 12166881
- [Background] Turner LA, Tecklenburg-Lund SL, Chapman RF, Stager JM, Wilhite DP, Mickleborough TD. Inspiratory muscle training lowers the oxygen cost of voluntary hyperpnea. J Appl Physiol (1985). 2012 Jan;112(1):127-34. doi: 10.1152/japplphysiol.00954.2011. Epub 2011 Oct 6. PMID 21979803
- [Derived] Al-Rammahi U, Soukka T, Malinen J, Happonen RP, Sovijarvi A, Anttalainen U. Effects of steam-assisted respiratory muscle training on sleep apnoea symptoms and pulmonary function in men and women: a pilot study. Sleep Breath. 2025 Sep 15;29(5):286. doi: 10.1007/s11325-025-03449-2. PMID 40952626